CLINICAL TRIAL: NCT06629311
Title: Study of Platelet Count Changes During the Use of Autotransfusion Device in Cardiac Surgery
Brief Title: Platelet and Autotransfusion Device in Cardiac Surgery
Acronym: PLAQ-SES
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9264
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Platelets; Autotransfusion Device
Keywords: Cardiac surgery; Autotransfusion device; Platelets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 32 Days
Biospecimen Retention: Samples Without DNA — Platelet-poor plasma Used autotransfusion device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Autotransfusion device — Standard cardiac surgery using I-SEP and SAME™ autotransfusion device

SUMMARY:
Cardiac surgery is a bleeding-risk surgery and frequently requires blood transfusion. Intraoperative autotransfusion devices are used to aspirate, process and retransfuse patients' blood. These devices are effective in recovering red blood cells and limiting the need for transfusion of packed red blood cells. Some devices, such as I-SEP's SAME®, can also be used to recover platelets, but their effectiveness has not yet been evaluated in real-life situations. The aim of this study is therefore to investigate the evolution of platelet counts following the use of an intraoperative recovery device in adult patients undergoing standard cardiac surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Having undergone standard cardiac surgery (excluding redux surgery, dissection, endocarditis, circulatory assist and transplants)
* Treated with an autotransfusion device during the surgery
* Subject having expressed their consent to the study

Exclusion Criteria:

* Anemia less than 7 g/dL
* Pregnant women
* Redux surgery, dissection, endocarditis, circulatory assistance, and transplants
* Contraindication to the use of an autotransfusion device
* Impossibility of giving the subject informed information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients addressed in a university hospital for cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2026-09-08 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Platelet count | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device
  Study the evolution of platelet counts following the use of I-SEP's SAME™ autotransfusion device in major patients undergoing standard cardiac surgery

SECONDARY OUTCOMES:
To study the evolution of platelet count following the use of the autotransfusion device (other than SAME) in major patients undergoing standard cardiac surgery. | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device
To study the evolution of platelet function (flow cytometry and flow aggregation) following the use of a autotransfusion device in major patients undergoing standard cardiac surgery. | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device
Study the evolution of platelet function according to the autotransfusion device used. | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device
Study post-operative bleeding volume as a function of autotransfusion device type. | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device
Study the volume of labile blood product transfusion according to the autotransfusion device used. | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device
Study the intensity of post-operative inflammatory syndrome as a function of the autotransfusion device used. | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device
Study platelet adhesion to the autotransfusion device membranes using electron microscopy. | Before the use of blood sparing system and 5 minutes after the end of the infusion of blood from the autotransfusion device

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: No